CLINICAL TRIAL: NCT04804293
Title: Treatment Monitoring of Carpal Tunnel Syndrome Using Shear Wave Elastography: A Pilot in Vivo Study
Brief Title: Assessment of Carpal Tunnel Syndrome by Shearwave Elastography
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Azra Alizad, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-001106
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Shear Wave Elastography; Peripheral compression neuropathy; Neuropathy; Demyelination
MeSH Terms: conditions — Carpal Tunnel Syndrome; Demyelinating Diseases

STUDY DESIGN:
Intervention Model Description: Central hypothesis is that SWE provides quantitative information about the physical properties of the MN and surrounding tissue that help to identify carpal tunnel syndrome, its severity and response to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Operative treatment (surgical decompression) for carpal tunnel syndrome (Experimental): Shear wave elastography (SWE) will be used to assess the stiffness of tissue. Patients will be revaluated at 3 and 6 months post-operatively. Patient will sit done in a chair. The investigators will scan the wrist area of both arms to acquire SWE map. This imaging will be done before the treatment. We will repeat the imaging study at 3 and 6 months after the treatment. Each ultrasound imaging session will take about less than 10 min. The investigators do not expect any discomfort during the imaging.
  Interventions: Device: FDA approved ultrasound system with shear wave elastography capability
- Corticosteroid injection treatment for carpal tunnel syndrome (Experimental): Shear wave elastography (SWE) will be used to assess the stiffness of tissue. Patients will be revaluated after 6 weeks following corticosteroid injection. Patient will sit done in a chair. The investigators will scan the wrist area of both arms to acquire SWE map. The investigators do not expect any discomfort during the imaging.
  Interventions: Device: FDA approved ultrasound system with shear wave elastography capability

INTERVENTIONS:
Device: FDA approved ultrasound system with shear wave elastography capability — The investigators will acquire at least 4 acquisitions for each of 2 locations on the wrist. The objective is to correlate SWE measurements with patient-reported measures of symptom severity and functional status scores and severity of pre-operative electrodiagnostic tests (EDX). Evaluate the treatment response to surgical decompression or corticosteroid injection, using quantitative SWE and correlate the results to repeated patient reported outcomes with Boston CTQ, and objective clinical improvement with Semmes-Weinstein monofilament evaluation for recovery of sensibility, and grip and lateral pinch strength.

SUMMARY:
This study is being done to test a new ultrasound method to detect possible stiffness problems within wrist(s). The purpose of this research is to the test the effectiveness of a new ultrasound method to check the nerve and surrounding tissue in both wrist of patient volunteers before and after treatment.

DETAILED DESCRIPTION:
The ultrasound system is FDA approved. The risks associated with this research study are not beyond the normal risk of conventional ultrasound and should not cause you any discomfort. Ultrasound at the intensity levels and duration used in this study has not been shown to present risk to humans. The investigators will conduct the SWE study on the set time point when the patient returns for follow-up after the therapy (surgical decompression or corticosteroid injection).

A set of pictures will be taken of patients wrists by the FDA approved ultrasound system. This system uses a special type of ultrasound for imaging your wrists.

The ultrasound study will be repeated after 3 and 6 months after the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers.
* Age ≥ 18 years old.
* Having unilateral symptom of wrist pain
* Scheduled for corticosteroid injection or surgery

Exclusion Criteria:

* Individuals less than 18 years of age.
* Prior surgery.
* People considered in "vulnerable" populations.
* Having bilateral symptoms

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the treatment response by shear wave elastography (SWE) | First 3 months
  Evaluate the treatment response to surgical decompression or corticosteroid injection, using quantitative SWE and correlate the results to repeated patient reported outcomes with Boston CTQ, and objective clinical improvement with Semmes-Weinstein monofilament evaluation for recovery of sensibility, and grip and lateral pinch strength.

SECONDARY OUTCOMES:
Correlate shear wave elastography (SWE) measurements with patient-reported measures of symptom severity and functional status scores and severity of pre-operative electrodiagnostic tests (EDX) elasticity | 3 to 6 months
  Determine the severity and patient outcome scores in patients with symptoms of CTS and Correlate the symptom severity and functional status assessed by the Boston Carpal tunnel Questionnaire (CTQ)21 validated patient outcome scoring profile) in patients with diagnosis of carpal tunnel syndrome with SWE determined median nerve (MN) stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No